CLINICAL TRIAL: NCT02565420
Title: Saline Versus Lactated Ringer's Solution: The SOLAR Fluid Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kamal Maheshwari, MD MPH, Principal Investigator, The Cleveland Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 15-858
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Saline Solution; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Alternating intervention
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactated Ringer's solution (Active Comparator): During the perioperative period of the colorectal, orthopedic or similar surgery the patient will receive an intervention of Lactated Ringer's solution fluids.
  Interventions: Other: Lactated Ringer's solution
- normal saline (Placebo Comparator): During the perioperative period of the colorectal, orthopedic or similar surgery the patient will receive an intervention of normal saline solution.
  Interventions: Other: Normal saline

INTERVENTIONS:
Other: Normal saline — Patients will be administered normal saline for intraoperative fluid management.
  Arms: normal saline
Other: Lactated Ringer's solution — Patients will be administered Lactated Ringer's solution for intraoperative fluid management.
  Arms: Lactated Ringer's solution

SUMMARY:
Perioperative volumes of saline cause a mild acidosis compared with buffered fluids. On the other hand, saline administration maintains plasma osmolality and better repletes vascular volume which is an important goal of perioperative fluid administration. Currently, there is no convincing evidence that either saline or buffered solutions are preferable. Consequently, both types of fluid remain in common use at the Clinic and worldwide.

There has never been a large trial of perioperative saline and balanced salt solutions comparing the incidence of major complications including acute kidney injury. The investigators primary objective is thus to determine the relative safety of perioperative saline and lactated Ringer's solution. Specifically, the investigators propose to test the:

1. Primary hypothesis that a composite of major in-hospital postoperative complications is lower in patients given lactated Ringer's solution compared to normal saline.
2. Secondary hypothesis that acute kidney injury, measured by AKIN criteria, is lower in patients given lactated Ringer's solution compared to normal saline.

The acquisition cost of saline and lactated Ringer's solutions is similar in the United States. (Curiously, buffered solutions are far more expensive than saline in Great Britain.) But to the extent that one fluid or the other provokes more complications, cost of care may be increased with that fluid selection. Cost may also be increased by the need for additional electrolyte monitoring and electrolyte replacement.

The investigators will therefore secondarily conduct an economic evaluation to determine the relative incremental hospital cost of each fluid. To the extent that one fluid or the other reduces cost (assuming similar complication rates), the Clinic will be able to reduce cost by specifying the appropriate fluid without impairing quality.

Evidence that one fluid or the other causes few complications would be a strong quality indicator that the Clinic should standardize perioperative fluid selection.

ELIGIBILITY:
Inclusion Criteria:

* Patients having colorectal or similar surgery
* Patients having orthopedic or similar surgery
* Patients 18 years and older

Exclusion Criteria:

* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8616 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Major Post Operative Complications | After surgery through hospital discharge
  Major complications include in-hospital mortality, renal (AKIN criteria 2+), respiratory, infectious, and hematological complications.

SECONDARY OUTCOMES:
Economic evaluation | After surgery through hospital discharge
  The evaluation will determine the incremental costs between the two interventions; uncomplicated care and care of complications, as well as a combined incremental cost.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, M.D., Study Chair — Chair, Outcomes Research
Locations (1):
- General Anesthesia, Anesthesia Institute, Cleveland, Ohio, United States